CLINICAL TRIAL: NCT02325466
Title: Comparative Efficacy of Ticagrelor Versus Aspirin on Blood Viscosity in Peripheral Artery Disease (PAD) Patients With Type 2 Diabetes (T2D)
Brief Title: Comparative Efficacy of Ticagrelor Versus Aspirin on Blood Viscosity in Peripheral Artery Disease Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Robert Rosenson, Professor Medicine, Cardiology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 13-1925
Record Dates: First submitted 2014-12-19; First posted 2014-12-25 (Estimated); Results first posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Artery Disease; Type 2 Diabetes
Keywords: Peripheral Artery Disease; Type 2 Diabetes; Blood Viscosity; Ticagrelor; Aspirin
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus, Type 2 | interventions — Aspirin; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aspirin/Ticagrelor placebo (Placebo Comparator): aspirin 81 mg daily and ticagrelor placebo twice daily
  Interventions: Drug: Aspirin; Drug: Ticagrelor Placebo
- Aspirin/Ticagrelor (Active Comparator): aspirin 81 mg daily and ticagrelor 90 mg twice daily
  Interventions: Drug: Aspirin; Drug: Ticagrelor
- Aspirin Placebo/Ticagrelor (Active Comparator): aspirin placebo daily and ticagrelor 90 mg twice daily
  Interventions: Drug: Ticagrelor; Drug: Aspirin Placebo

INTERVENTIONS:
Drug: Aspirin — Aspirin 81mg
  Other Names: ASA
  Arms: Aspirin/Ticagrelor; Aspirin/Ticagrelor placebo
Drug: Ticagrelor — ticagrelor 90 mg
  Arms: Aspirin Placebo/Ticagrelor; Aspirin/Ticagrelor
Drug: Aspirin Placebo
  Other Names: Placebo
  Arms: Aspirin Placebo/Ticagrelor
Drug: Ticagrelor Placebo
  Other Names: Placebo
  Arms: Aspirin/Ticagrelor placebo

SUMMARY:
The hypothesis being that both aspirin-ticagrelor and ticagrelor monotherapy will be superior to aspirin monotherapy in the reduction of whole blood viscosity at the end of each 4 week treatment period. Study participants will be randomized into 3 groups, and each group will receive each of 3 treatments in the cross-over study. At the end of each individual 4 week treatment period the investigators will determine whether there are differences in low and high shear rate dependent viscosity and investigate the effect of the treatment on peripheral arterial blood flow using pulse volume recordings, ankle brachial index and toe pressures. Subjects will be eligible if they have ankle-brachial index less than or equal to 0.85, or if a patient's blood vessels are calcified, patients will have toe-brachial index less than or equal to 0.6 performed using continuous-wave Doppler.

DETAILED DESCRIPTION:
Ticagrelor has been shown to significantly reduce the rate of cardiovascular disease (CVD) events and death compared with clopidogrel in patients having prior acute coronary syndrome. A number of outcome studies have demonstrated the risk of major CVD events increased with blood viscosity. Stroke patients and those with stroke risk factors were shown to have chronically elevated blood viscosity relative to healthy controls. Based on prior observations, the rationale for this study is to demonstrate that both aspirin-ticagrelor and ticagrelor monotherapy will be superior to aspirin monotherapy in the reduction of whole blood viscosity at the end of each 4 week treatment period.

The primary objectives for this study is to: (1) Compare the effect of aspirin-ticagrelor with aspirin in a double blind, randomized, cross-over study design (weeks 1-4, weeks 6-10, and weeks 12-16) on blood viscosity at both low (5 s-¹) and high (300 s-¹) shear rates at the end of each 4-week treatment period; and (2) to compare the effect of ticagrelor mono-therapy with aspirin in a double blind, randomized, cross-over study design (weeks 1-4, weeks 6-10, and weeks 12-16) on blood viscosity at both low (5 s-¹) and high (300 s-¹) at the end of each 4-week treatment.

The secondary objectives for this study include: (1) a determination as to whether there are differences in low and high shear rate dependent viscosity with treatment by ticagrelor alone and combination aspirin-ticagrelor. Additionally, investigated will be the effect of the treatment on peripheral arterial blood flow using pulse volume recordings, ankle brachial index, and toe pressures.

The general approach to evaluation of drug efficacy will be through blood samples collected with a standard venipuncture for viscosity testing. Blood viscosity will be measured using an automated scanning capillary tube viscometer across a physiologic range of shear rates of 1-1000 s-1 in increments of 0.1 s-1. Blood viscosity levels at 5 s-1 will be reported as low-shear viscosity, and blood viscosity measurements at 300 s-1 will be reported as high-shear viscosity. Additionally, pulse volume recordings will be simultaneously obtained at the level of the ankle, metatarsal and toe bilaterally according to standard protocol, and Continuous-wave Doppler will be used to determine ankle-brachial indices or toe-brachial indices, and flow velocity profiles.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged ≥ 35 years
* Type 2 diabetes mellitus
* Symptomatic PAD
* Ankle-brachial index ≤ 0.85 or calcified blood vessels with toe-brachial index ≤ 0.6 and/or abnormal post-exercise ankle-brachial index
* Prior surgical or percutaneous intervention of the peripheral arteries ≥12 months previously with a residual stenoses of ≥50% in a non-dilated artery.

Exclusion Criteria:

* Subject is pregnant or breast-feeding
* Planned revascularization or amputation
* Known bleeding disorder
* History of intracranial hemorrhag3
* Considered at risk of hemorrhagic events
* Hypersensitivity or allergic reactions to aspirin
* Concomitant use of anticoagulants such as warfarin, dabigatran, factor Xa inhibitors or antiplatelet drugs such as clopidogrel, dipyridamole and sulfapyridine
* Subject has a condition or circumstance which would prevent them from adhering to treatment regimens
* Subject has active infection
* Subject has an anemia
* Subject has given blood or received a blood transfusion at any point during the study
* Subject has polycythemia vera or any hyperviscosity syndrome
* Subjects with Waldenstrom's macroglobulinemia who have an increased risk of hyperviscosity syndrome
* Subject has history of severe liver disease, obstructive liver disease such as primary biliary cirrhosis or end-stage renal disease (eGFR <30 mL/min/m2)
* Family members or employees of the investigator or study centers involved in the study
* Subject has poor diabetes or hypertension control (systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 100 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-04; Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rosenson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Rosenson RS, Chen Q, Najera SD, Krishnan P, Lee ML, Cho DJ. Ticagrelor improves blood viscosity-dependent microcirculatory flow in patients with lower extremity arterial disease: the Hema-kinesis clinical trial. Cardiovasc Diabetol. 2019 Jun 7;18(1):77. doi: 10.1186/s12933-019-0882-5. PMID 31174526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from April 2015 to April 2018. Study participants were recruited from the outpatient cardiology practice and the Cardiac Catheterization database at the Mount Sinai Hospital, New York, NY, USA.
Groups:
- Aspirin/Ticagrelor Placebo: aspirin 81 mg daily and ticagrelor placebo twice daily
  crossover order was never unblinded to PI and study team
- Aspirin/Ticagrelor: aspirin 81 mg daily and ticagrelor 90 mg twice daily
  crossover order was never unblinded to PI and study team
- Aspirin Placebo/Ticagrelor: aspirin placebo daily and ticagrelor 90 mg twice daily
  crossover order was never unblinded to PI and study team
Period: Period 1 Timeframe - Baseline to Week 4
Arm/Group | Aspirin/Ticagrelor Placebo | Aspirin/Ticagrelor | Aspirin Placebo/Ticagrelor
Started | 23 | 23 | 24
Completed | 22 | 21 | 21
Not Completed | 1 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — urgent vascularization | 1 | 0 | 2
Period: Period 2 - Timeframe Week 4 to Week 10
Arm/Group | Aspirin/Ticagrelor Placebo | Aspirin/Ticagrelor | Aspirin Placebo/Ticagrelor
Started | 22 | 21 | 21
Completed | 19 | 20 | 21
Not Completed | 3 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — urgent vascularization | 1 | 0 | 0
Period: 3rd Crossover - Week 10 to Week 16
Arm/Group | Aspirin/Ticagrelor Placebo | Aspirin/Ticagrelor | Aspirin Placebo/Ticagrelor
Started | 19 | 20 | 21
Completed | 18 | 18 | 21
Not Completed | 1 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — urgent vascularization | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Two crossovers with all participants experiencing all 3 arms
Arm/Group | All Participants
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 23
  More than one race | 21
  Unknown or Not Reported | 0
Hematocrit [Mean (Standard Deviation); unit: percent of cells] | 38.3 (4.4)
Fibrinogen [Mean (Standard Deviation); unit: mg/dL] | 351 (109)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 124 (47)
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of hemoglobin] | 7.20 (1.1)
Blood viscosity 300 s^-1 [Mean (Standard Deviation); unit: centipoises (cPs)] — Blood viscosity is a measure of the resistance of blood to flow. Blood viscosity measured at a shear rate of 300 s^-1
  centipoises (cPs) | 4.0 (0.6)
Blood viscosity 5 s^-1 [Mean (Standard Deviation); unit: cPs] — Blood viscosity measured at a shear rate of 5 s^-1
  cPs | 11.1 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Low Shear Blood Viscosity
Description: Compare the effect of aspirin-ticagrelor and ticagrelor monotherapy with aspirin on blood viscosity from week 16 to baseline
Time Frame: baseline, week 16
Population: data collected and included for any participants who return for any of their visits.
Measure: Mean (Standard Deviation); unit: 5 s^-1 cPs
Arm/Group | Aspirin/Ticagrelor Placebo | Aspirin/Ticagrelor | Aspirin Placebo/Ticagrelor
Number analyzed (Participants) | 60 | 61 | 58
5 s^-1 cPs | 1.045 (1.525) | -1.793 (1.835) | -1.759 (1.298)

2. Primary Outcome: Mean Change in High Shear Blood Viscosity
Description: Compare the effect of aspirin-ticagrelor and ticagrelor monotherapy with aspirin on blood viscosity at week 16 to baseline
Time Frame: baseline and week 16
Population: data collected and included for any participants who return for any of their visits.
Measure: Mean (Standard Deviation); unit: 300 s^-1 cPs
Arm/Group | Aspirin/Ticagrelor Placebo | Aspirin/Ticagrelor | Aspirin Placebo/Ticagrelor
Number analyzed (Participants) | 60 | 61 | 58
300 s^-1 cPs | 0.165 (0.318) | -0.228 (0.469) | -0.231 (0.360)

3. Secondary Outcome: Mean Change in Peripheral Arterial Blood Flow
Description: Measure of treatment effect using pulse volume recordings of the ankle, great toe and brachial artery to calculate the ankle brachial index (ABI) and toe brachial index (TBI) at week 16 compared to baseline.
  ABI and TBI are taken in order to determine the existence and severity of peripheral arterial disease.
  ABI - The normal range for the ankle-brachial index is between 0.90 and 1.30. ABI <0.90 is abnormal: 0.41 to 0.90 indicates mild to moderate peripheral artery disease; 0.40 and lower indicates severe disease. The lower the index, the higher the chances of leg pain while exercising or limb-threatening low blood flow.
  TBI ≥ 0.7 is normal, TBI < 0.7 is abnormal.
Time Frame: baseline and week 16
Population: data collected for participants who return for their visits.
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Aspirin/Ticagrelor Placebo | Aspirin/Ticagrelor | Aspirin Placebo/Ticagrelor
Number analyzed (Participants) | 60 | 61 | 58
index
  ABI right side | 0.038 (0.055) | 0.021 (0.019) | 0.095 (0.051)
  ABI left side | 0.015 (0.067) | 0.032 (0.038) | 0.075 (0.029)
  TBI right side | 0.044 (0.013) | 0.009 (0.015) | 0.011 (0.008)
  TBI left side | 0.004 (0.022) | -0.016 (0.018) | 0.036 (0.028)

4. Secondary Outcome: Mean Change in Microvascular Blood Flow Composite Score
Description: Measure of treatment effect using pulse volume recordings of the ankle, great toe and brachial artery to calculate the ankle brachial index and toe pressures composite score at week 16 from baseline. Composite score obtained by adding all the measurements and averaged. The score was tested by the Laser Doppler Flowmetry (LDF). Minimum score is 0 which mean no blood flow detected and there is no maximum value of the score, and higher score mean better blood flow.
Time Frame: baseline and week 16
Population: data collected for participants who return for their visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aspirin/Ticagrelor Placebo | Aspirin/Ticagrelor | Aspirin Placebo/Ticagrelor
Number analyzed (Participants) | 60 | 61 | 58
score on a scale
  Right side | -4.10 (13.30) | 13.64 (7.34) | -5.23 (7.76)
  Left side | -5.60 (11.86) | 24.76 (8.36) | -4.29 (7.48)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: data collected for participants who return for any subsequent visits
Arm/Group | Aspirin/Ticagrelor Placebo | Aspirin/Ticagrelor | Aspirin Placebo/Ticagrelor
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 1/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70 | 1/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin/Ticagrelor Placebo (N=70) | Aspirin/Ticagrelor (N=70) | Aspirin Placebo/Ticagrelor (N=70)
GI Bleeding (Gastrointestinal disorders) | 0 | 1 | 0 — prolonged hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin/Ticagrelor Placebo (N=70) | Aspirin/Ticagrelor (N=70) | Aspirin Placebo/Ticagrelor (N=70)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT02325466/Prot_SAP_000.pdf